CLINICAL TRIAL: NCT01506817
Title: Dynamic Contrast Enhanced MRI of the Hands in Patients With Fibromyalgia. A Pilot Study
Brief Title: Dynamic Contrast Enhanced (DCE)-MRI in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Oak Foundation (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, MD, DMSci, Frederiksberg University Hospital
Other Study IDs: HB-030112
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; DCE-MRI; neurogenic inflammation; contrast-enhancement patterns
MeSH Terms: conditions — Fibromyalgia; Neurogenic Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Fibromyalgia: patients with fibromyalgia fulfilling the 1990-ACR research criteria and with pain in the hands as a prominent clinical feature
  Interventions: Procedure: Dynamic contrast-enhanced MRI of the hands
- Controls: healthy aged matched pain-free controls
  Interventions: Procedure: Dynamic contrast-enhanced MRI of the hands

INTERVENTIONS:
Procedure: Dynamic contrast-enhanced MRI of the hands — The hand and wrist will be examined in a 3T Siemens Verio® MR scanner with the patients and normal controls supine and the hand along the side of the body (3T Verio) using a semiflex 15 channel body coil. Total imaging time varies between 30-35 minutes.

SUMMARY:
The primary objective of the current pilot study is to analyze MRI contrast-enhancement patterns in the hands of patients with fibromyalgia as compared to the findings in healthy controls. Further, to compare enhancement patterns obtained in fibromyalgia patients with those described in inflammatory joint disorders, i.e. rheumatoid arthritis and psoriatic arthritis.

Hypothesis:

Dynamic contrast-enhanced MRI (DCE-MRI) of the hands in patients with fibromyalgia reveals pathological imaging patterns indicative of diffuse non-arthrogenic inflammation of e.g. superficial soft tissues and /or muscle with patterns distinct from those of inflammatory joint disorders e.g. rheumatoid arthritis and psoriatic arthritis.

DETAILED DESCRIPTION:
Systematic, diagnostic studies applying DCE-MRI have never been performed in patients with fibromyalgia. However, characteristic contrast-enhancement patterns different from those seen in patients with rheumatoid arthritis and psoriatic arthritis have been observed in a small sample of fibromyalgia patients referred for DCE-MRI of the hands for differential diagnostic purposes at department of radiology, Frederiksberg Hospital. In these patients enhancement parameters indicative of vasodilatation and diffuse hyperperfusion involving subcutaneous tissues and muscles of the hands and fingers were found, whereas no synovial inflammation in joints or tendons could be demonstrated in the majority of these patients. Whether these observations are part of a "normal" physiological perfusion in healthy individual or a potential novel marker of disease activity remains to be studied.

If a pathological imaging pattern indicative of superficial soft tissue or muscle inflammation/hyper perfusion can be demonstrated it will have far-reaching implications for future research related to this patient population. Not only may this line of research contribute to a better neurobiological understanding of fibromyalgia and the neurobiological link between inflammation and pain modulation, but also to the development of more objective examination methods, which will make diagnosing more reliable and less subjective. Further, a better understanding of the neurobiology and phenomenological manifestations of fibromyalgia may have critical treatment implications

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Fibromyalgia according to the 1990-ACR research criteria
* Pain in the hands as a prominent clinical feature

Exclusion Criteria:

* Other know medical condition capable of causing patients symptoms (e.g. uncontrolled inflammatory/autoimmune disorder, uncontrolled endocrine disorder, malignancy)
* Renal impairment
* Contraindications for MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia recruited from Department of Rheumatology, Frederiksberg Hospital. Inclusion in the study will be based on clinical assessment by a specialist in rheumatology and member of the research team. Patients fulfilling the 1990-ACR criteria for fibromyalgia and with pain in the hands as a prominent clinical feature will be referred for DCE-MRI as part of the diagnostic workup.
  Healthy controls will be recruited by advertisement at www.forsøgsperson.dk or in the daily press and included in the project based on written, informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Imaging patterns obtained at DCE-MRI using the software program DYNAMIKA (www.imageanalysis.org.uk) of the dominant hand as evaluated by a specialist in radiology will be the primary outcome of the study. | at baseline
  The hand and wrist will be examined in a 3T Siemens Verio® MR scanner with the patients and normal controls supine and the hand along the side of the body (3T Verio) using a semiflex 15 channel body coil.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Boesen, MD,PhD, Principal Investigator — The Parker Institute and Department of Radiology, Frederiksberg Hospital Denmark; Henning Bliddal, Professor, DMSci, Study Director — The Parker Institute, Frederiksberg Hospital Denmark; Kirstine Amris, MD, Principal Investigator — The Parker Institute and Department of Rheumatology, Frederiksberg Hospital Denmark; Peter Taylor, Professor, MA, PhD, Principal Investigator — Kennedy Institute of Rheumatology, University of Oxford, England
Locations (1):
- The Parker Institute, Frederiksberg University Hospital, Frederiksberg, Denmark

REFERENCES:
- See also: Related Info — http://www.frederiksberghospital.dk/parker